CLINICAL TRIAL: NCT02727335
Title: Description of Clinical Anatomical Features and Long Term Follow-up for Patients With ALK Rearrangements
Acronym: CLINALK
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Other Study IDs: IFCT-1302
Record Dates: First submitted 2016-03-09; First posted 2016-04-04 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Non-small Cell Lung Cancer; Anaplastic Lymphoma Kinase Gene Mutation
Keywords: Non-squamous non-small cell lung cancer; crizotinib; real-world study; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients ALK + who received crizotinib: patients with ALK rearrangement who started treatment with crizotinib (250 mg twice a day) between the 18/11/2010 and the 31/12/2013 (will include patients from the ATU programs and patients treated after the marketing of crizotinib)

SUMMARY:
Description of clinical and anatomical features and long-term follow-up for patients with ALK rearrangement and treated by crizotinib

DETAILED DESCRIPTION:
Several French studies on crizotinib have been conducted in recent years. These are not only patients treated in the PROFILE 1005 and 1007 clinical studies but also patients who have been treated with crizotinib in the named patient ATU followed by the cohort ATU (Expended Access Cohort). Under the ATU program and according to ATU regulations, a limited set of data is collected and furthermore the follow up is stopped as soon as the ATU program closes. Thus it is not possible to have access to long term data and post progression data. Our project is to collect data from the patients from the ATU program (named patient and cohort) and if possible patients treated after the marketing of crizotinib, before, during and after crizotinib therapy. Centers selected for this observational study will be those of the IFCT network that took part in the ATU program.

This will allow an accurate analysis of crizotinib therapy under "real life" conditions. It should be emphasized that this information is generally neither available from clinical trials nor from ATU programs.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have locally advanced or metastatic NSCLC (Stage IIIb or Stage IV by AJCC 7th.) with positive ALK determined by IHC and/or FISH.
* Patient who received crizotinib on an expanded access basis (compassionate use) (ATU) due to their inability to meet eligibility criteria for on-going recruiting trials, inability to participate in other clinical trials (e.g., poor performance status, lack of geographic proximity), or because other medical interventions are not considered appropriate or acceptable
* Patient who received marketed crizotinib as a result of the standard care of metastatic NSCLC (Stage IIIb or Stage IV by AJCC 7th.) with positive ALK will also be eligible.
* Patient was able to swallow capsules and had no surgical or anatomical condition that precluded the patient from swallowing and absorbing oral medications on an ongoing basis.
* Patient has taken at least 1 week of treatment

Exclusion Criteria:

* Patient included in a crizotinib clinical trial
* Patient with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC carrying the ALK rearrangement in the named patient or cohort crizotinib ATU. This will be supplemented, where possible, by the patients with crizotinib prescriptions under the Marketing Authorisation.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  overall survival post-progression on crizotinib

SECONDARY OUTCOMES:
rare and severe complications of crizotinib therapy | 5 years
  Incidence of rare and severe complications of crizotinib therapy: hepatotoxicity, interstitial pneumonitis, diastolic heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Denis Moro-Sibilot, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique; Michael Duruisseaux, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (63):
- France (63):
  - Agen - CH, Agen
  - Angers - CHU, Angers
  - Angoulême - CH, Angoulême
  - Annecy - CH, Annecy
  - Avignon - Institut Sainte-Catherine, Avignon
  - CHU Besancon - Pneumologie, Besançon
  - Bordeaux - Clinique Saint Augustin, Bordeaux
  - Boulogne - Hôpital Ambroise Paré, Boulogne
  - Brest - Hôpital du Morvan, Brest
  - CH de Cannes, Cannes
  - CH Chambery, Chambéry
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Clermont-Ferrand - Centre Jean Perrin, Clermont-Ferrand
  - Colmar - CH, Colmar
  - CH de Dax, Dax
  - Dijon - CHU, Dijon
  - Dole - Centre Hospitalier Louis Pasteur, Dole
  - Douai - CH, Douai
  - Fréjus - CHI Saint Raphaël, Fréjus
  - Grenoble - Institut Daniel Hollard, Grenoble
  - CHRU Grenoble, Grenoble
  - Centre Hospitalier - Pneumologie, Le Havre
  - Centre Hospitalier - Pneumologie, Le Mans
  - Libourne - CH, Libourne
  - Centre Oscar Lambret, Lille
  - Limoges - Hôpital du Cluzeau, Limoges
  - Longjumeau - CH, Longjumeau
  - Marseille - Hôpital Saint Joseph, Marseille
  - Marseille - CRLCC, Marseille
  - Polyclinique du Parc, Maubeuge
  - Mâcon - CH, Mâcon
  - Meaux - CH, Meaux
  - Meulan - CHI, Meulan-en-Yvelines
  - CH de Mulhouse, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - Paris - Hôpital Cochin, Paris
  - Paris - Hôpital Saint Joseph, Paris
  - Paris - Hôpital Européen Georges Pompidou, Paris
  - Hopital Tenon - Pneumologie, Paris
  - Paris - Curie, Paris
  - Pau - CH, Pau
  - Lyon Sud, Pierre-Bénite
  - CHU, Poitiers
  - Reims - Institut Courlancy, Reims
  - Rennes - Clinique Saint Laurent, Rennes
  - Rodez - CH, Rodez
  - Rouen - CHU, Rouen
  - Saint Denis de la Réunion - CHD Guyon, Saint-Denis
  - Saint Herblain - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain
  - Saint-Julien-en-Genvois - CHI, Saint-Julien-en-Genevois
  - Saint Priest en Jarez - ICL, Saint-Priest-en-Jarez
  - Strasbourg - NHC, Strasbourg
  - Strasbourg - Centre Paul Strauss, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Centre Hospitalier Intercommunal, Toulon
  - Toulouse - Clinique Pasteur, Toulouse
  - Toulouse - CHU Larrey, Toulouse
  - Tours - CHU, Tours
  - Troyes - CH, Troyes
  - Vannes - Centre Hospitalier Bretagne Atlantique, Vannes
  - Vénissieux - Groupe Hospitalier Mutualiste les Portes du Sud, Vénissieux
  - CH de Villefranche - Pneumologie, Villefranche
  - Villejuif - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duruisseaux M, Besse B, Cadranel J, Perol M, Mennecier B, Bigay-Game L, Descourt R, Dansin E, Audigier-Valette C, Moreau L, Hureaux J, Veillon R, Otto J, Madroszyk-Flandin A, Cortot A, Guichard F, Boudou-Rouquette P, Langlais A, Missy P, Morin F, Moro-Sibilot D. Overall survival with crizotinib and next-generation ALK inhibitors in ALK-positive non-small-cell lung cancer (IFCT-1302 CLINALK): a French nationwide cohort retrospective study. Oncotarget. 2017 Mar 28;8(13):21903-21917. doi: 10.18632/oncotarget.15746. PMID 28423535
- See also: Official website — http://www.ifct.fr